CLINICAL TRIAL: NCT00540800
Title: Phase III Multicenter Study of the Effects on Quality of Life of Three-weekly Versus Weekly First-line Chemotherapy for Metastatic or Locally Advanced Breast Cancer
Brief Title: BREAST-10: Three-weekly Versus Weekly First-line Chemotherapy for Metastatic or Locally Advanced Breast Cancer
Acronym: BREAST-10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BREAST-10
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: anthracycline pre-treated; chemotherapy; first-line; metastatic breast cancer; locally advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Epirubicin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Three-weekly chemotherapy
  Interventions: Drug: docetaxel; Drug: epirubicin; Drug: capecitabine
- B (Experimental): Weekly chemotherapy
  Interventions: Drug: docetaxel; Drug: epirubicin; Drug: capecitabine

INTERVENTIONS:
Drug: docetaxel — given in combination with epirubicin or capecitabine
Drug: epirubicin — for patients with locally advanced breast cancer, or metastatic breast cancer not previously treated with anthracyclines
Drug: capecitabine — for metastatic breast cancer patients previously treated with anthracyclines

SUMMARY:
Some chemotherapies, including docetaxel, are better tolerated and just as effective when giving the dose weekly rather than on an every three week basis. The purpose of this study is to compare 2 schedules of combination chemotherapy with docetaxel for the effects on quality of life. Standard every three week chemotherapy will be compared with weekly chemotherapy for metastatic or locally advanced breast cancer.

DETAILED DESCRIPTION:
Patients with locally advanced breast cancer and patients with metastatic breast cancer who have not previously received an anthracycline will be treated with docetaxel and epirubicin.

Patients with metastatic breast cancer who have already received anthracyclines will be treated with docetaxel and capecitabine.

All patients will be randomized to receive their treatment either on an every three week schedule, or on a weekly schedule.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of breast cancer
* Inoperable locally advanced or metastatic disease not yet treated with first-line chemotherapy
* Age < 70 years
* ECOG performance status < 2
* Written informed consent

Exclusion Criteria:

* Previous or concomitant malignant neoplasm (excluding adequately treated baso or spinocellular skin carcinoma or carcinoma in situ of the cervix)
* Previous treatment with docetaxel
* Symptomatic brain metastases
* Neutrophil < 2000/mm3, platelets < 100,000/mm3, haemoglobin < 10 g/dl
* Creatinine > 1.25 x the upper normal limits
* GOT and/or GPT > 1.25 x the upper normal limits in absence of hepatic metastases
* GOT and/or GPT > 2.5 x the upper normal limits in presence of hepatic metastases
* Bilirubin > 1.5 x the upper normal limit
* Any concomitant pathology that would, in the investigator's opinion, contraindicate the use of the drugs in this study
* Inability to provide informed consent
* Inability to comply with follow-up

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2004-02; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
quality of life | during first 6 weeks of chemotherapy

SECONDARY OUTCOMES:
Response rate | After 12 and 24 weeks of chemotherapy
Toxicity | every 3 weeks
overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea de Matteis, M.D., Principal Investigator — NCI Naples, Division of Medical Oncology C; Francesco Perrone, M.D., Ph.D., Principal Investigator — NCI Naples, Clinical Trials Office
Locations (3):
- Italy (3):
  - Istituto Nazionale dei Tumori , Divisione di Oncologia Medica B, Napoli
  - Istituto Nazionale dei Tumori, Divisione di Oncologia Medica C, Napoli
  - Ospedale S. Luca ASL SA 3, Vallo della Lucania

REFERENCES:
- [Result] Nuzzo F, Morabito A, Gravina A, Di Rella F, Landi G, Pacilio C, Labonia V, Rossi E, De Maio E, Piccirillo MC, D'Aiuto G, Thomas R, Rinaldo M, Botti G, Di Bonito M, Di Maio M, Gallo C, Perrone F, de Matteis A. Effects on quality of life of weekly docetaxel-based chemotherapy in patients with locally advanced or metastatic breast cancer: results of a single-centre randomized phase 3 trial. BMC Cancer. 2011 Feb 16;11:75. doi: 10.1186/1471-2407-11-75. PMID 21324184